CLINICAL TRIAL: NCT03948204
Title: Socioeconomic Status, Differences in Quality of Life and Shared Decision Making Among Patients With Non-metastatic Prostate Cancer
Brief Title: Quality of Life and Shared Decision Making in Prostate Cancer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Norwegian Institute of Public Health (Other Government)
Responsible Party: Principal Investigator, Tom Børge Johannesen, Junior Head, Registry Dept, Norwegian Institute of Public Health
Other Study IDs: 0910
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prostate cancer: Men diagnosed with prostate cancer
- Men without prostate cancer: Men without prostate cancer matched for age and county

SUMMARY:
"Life after prostate cancer" is a prospective, population-based, case-control study where all men diagnosed with Prostate cancer (PCa) from 01.01.2017 regardless of age and disease stage are invited to a survey by questionnaire on their health. Men with no history of PCa are identified through the National Registry, matched on age and region of residence, and invited to the survey as controls. Patients and controls who have signed up for an official digital mailbox are invited electronically. Those who do not have a digital mailbox are invited by regular mail. All participants have given their informed consent for all linkages planned in this study. Due to electronic reporting of histological reports to the Norwegian Prostate Cancer Registry, patients are invited to the survey shortly after diagnosis. More than 6 400 patients have submitted questionnaires per April 2019.

DETAILED DESCRIPTION:
Survey participants complete questionnaires on adverse effects / functional outcomes and QoL. The survey questionnaire includes EQ-5D-5L and EORTC QLQ-C3). EPIC-26 is used together with additional questions on sexual interest and use of aids. Highest level of education, height, weight and marital status are also included at baseline. All those with PCa, as well as the men without PCa who participate at baseline, are invited to submit follow-up questionnaires 1 and 3 years after diagnosis. The same instruments are then used with the addition of questions on work ability together with questions on treatment and experience with the health care service including shared decision making. From Statistics Norway data on personal and household income will be available together with education level stated by participants. The Norwegian Prostate Cancer Registry, a national quality registry on PCa, is incorporated in The Cancer Registry of Norway and is in collaboration with clinical specialists from hospitals in all regions of the country. The registry publishes results regularly to patients and hospitals with updated statistics on incidence, work-up, treatment choice and outcomes. All variables concerning work-up, diagnosis (histopathological data, imaging) stage (cTNM, PSA, Gleason score), treatment (surgery, radiotherapy, endocrine treatment) and follow-up are available for linkage with questionnaire data from the patients. Patients will be stratified into low-, intermediate-, and high-risk groups as defined by the European Association of Urology based on the clinical T-category (cT), the PSA level, and the Gleason score (GS) at the time of diagnosis. Low-risk: cT1-T2a and PSA<10 ng/mL and GS<7, Intermediate-risk: cT2b or PSA 10-20 ng/ml or GS=7, high-risk localised: cT2c or PSA>20 ng/mL or GS>7, high-risk locally advanced: cT3-4 or cN1. Division will further be by initial treatment: radical prostatectomy, radiotherapy ≥74 Gy by standard fractionation with or without hormone treatment, or no local treatment consisting of active surveillance or watchful waiting. The Norwegian Patient Registry contains data on all individuals waiting for treatment or that have received treatment including both in- and outpatient specialist care. A modified version of the Charlson's comorbidity index shown to be valid for patient registry data will for this study be used.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with prostate cancer in Norway at or after 01.01.2017

Exclusion Criteria:

-

Ages: 0 Years to 110 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All men with prostate cancer in Norway
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Qality of life Global health status | 3 years
  Global health status from QLQ-C30 version 3.0 scale
Qality of life Physical functioning | 3 years
  Physical functioning from QLQ-C30 version 3.0 scale
Qality of life Role functioning | 3 years
  Role functioning from QLQ-C30 version 3.0 scale
Qality of life Emotional functioning | 3 years
  Emotional functioning from QLQ-C30 version 3.0 scale
Qality of life Cognitive functioning | 3 years
  Cognitive functioning from QLQ-C30 version 3.0 scale
Qality of life Social functioning | 3 years
  Social functioning from QLQ-C30 version 3.0 scale

CONTACTS AND LOCATIONS:
Locations (1):
- The Cancer Registy of Norway, Oslo, Norway